CLINICAL TRIAL: NCT00368602
Title: Beta Adrenergic Receptor Modulation of Burn Wound Healing
Brief Title: Beta Blocker for Chronic Wound Healing
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-06-00351
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Ulcer; Burns
MeSH Terms: conditions — Ulcer; Burns | interventions — Timolol; Adrenergic beta-Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): This group receives topical beta adrenergic antagonists (Timoptic) plus standard of care.
  Interventions: Drug: Timoptic
- 2 (Placebo Comparator): The group will be given standard of care with placebo medication.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Timoptic — Timoptic to be applied to the target wound daily for up to 12 weeks.
  Other Names: beta adrenergic antagonists
  Arms: 1
Other: Placebo — Saline solution with no active ingredients to be applied to the target wound daily for up to 12 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of treatment of chronic cutaneous ulcers and burn wounds with topical beta adrenergic antagonists (Timoptic®).

DETAILED DESCRIPTION:
The purpose of this study is to learn more about how to heal venous leg ulcers faster and to test the safety of a drug and see what effects it has on a venous leg ulcer.

You will:

* be interviewed and examined
* have a physical exam
* have blood and urine tested
* have photographs taken of the wound
* apply medication to the leg ulcer as directed

ELIGIBILITY:
Inclusion Criteria:

* Any race btwn 18 and 85 years of age, inclusive;
* Male or female, neither pregnant nor lactating.
* Informed consent;
* Have at least 1 lower extremity ulcer in the gaiter area (knee to ankle):

  1. Surface area of ≥2 sq. cm. to ≤20 sq. cm.; Ulcer with largest surface area meeting inclusion criteria will be selected.
  2. If 2 ulcers present with the same surface area, ulcer of longest duration selected.
  3. Study ulcer must be at least 2 cm from any other ulcer on same extremity.
  4. A viable wound bed free of necrotic tissue post-debridement, if debridement is indicated.

     5. Have an Ankle Brachial Index (ABI) >0.7; 6. Presence of either dorsalis pedis or posterior tibialis pulses by Doppler on the study extremity; 7. Have a non-healing (open) ulcer for at least 1 month. Subjects who failed conservative therapy are eligible for the study; 8. Comply with a trial (13 to 17 days) of protocol-specified standard care prior to randomization; 9. Two or more of the following: dermatitis, atrophie blanche, varicosities, hyperpigmentation or lipodermatosclerosis;

     Exclusion Criteria:
* Decrease in wound surface area of >35% btwn Screening and Visit 1 (Randomization);
* Cellulitis, osteomyelitis, ulcer with exposed bone, tendon or fascia, or purulent exudates in ulcer area;
* Grade IV ulcer;
* Evidence of study ulcer infection;
* Study ulcer of non-venous etiology;
* Acquired or are known to be infected with HIV;
* Uncontrolled diabetes mellitus;
* Immunodeficiency as defined by serum IgG, IgA, and IgM less than one-half the lower limit of normal;
* Severe protein malnutrition as defined by serum albumin <2.5 g/dL;
* Severe anemia defined as a total of hemoglobin of <10 g/dL for males or <8 g/dL for females;
* Chronic renal insufficiency requiring dialysis;
* Serum aspartate aminotransferase (AST, SGOT, GOT) or serum alanine aminotransferase (ALT, SGPT, GPT) levels greater than twice the upper limit of normal;
* New York Heart Association Functional Classification of IV;
* Deep vein thrombosis (DVT) w/in last 6 weeks or clinical evidence of current DVT;
* Arterial revascularization of the study extremity w/in previous 6 months from the date of Screening Visit;
* History, w/in previous 12 months from date of Screen Visit, of alcohol or drug abuse, particularly methadone or heroin;
* Received previous treatment with the following during the 60 days prior to Screening: Immunosuppressive agents, radiation, chemotherapy, growth factors at the site of the study ulcer, split- or full-thickness skin graft at the site of the study ulcer, biologically-active cellular or acellular product(s) at the site of the study ulcer, investigational drug or device
* Received previous treatment with systemic corticosteroids prior to Screening (Chronic corticosteroids w/in 90 days or short course corticosteroids w/in 30 days)
* Been hospitalized for treatment of any venous ulcer w/in the previous 30 days from Screening.
* Asthma or a history of asthma, obstructive pulmonary disease, myasthenia gravis, hyperthyroidism, history of heart block

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter will be complete ulcer healing, which is defined as 100% epithelialization with no drainage or need for an absorptive dressing. | 12 weeks

SECONDARY OUTCOMES:
100% re-epithelialization will be clinically determined at each visit by the Investigator. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rivkah R Isseroff, MD, Principal Investigator — University of California, Davis
Locations (1):
- VA Medical Center, Mather, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical/index.html